CLINICAL TRIAL: NCT02453685
Title: A 32-week Randomised, Multinational, Treat-to-target, Open Label, Parallel Group Comparison of Stepwise Insulin Intensification of Biphasic Insulin Aspart (BIAsp) 30 and Basal-bolus Therapy With Insulin Glargine and Insulin Aspart in Insulin naïve Type 2 Diabetic Patients Inadequately Controlled on Oral Anti-diabetic Therapy
Brief Title: A Study to Compare Insulin Intensification of Biphasic Insulin Aspart 30 and Insulin Analogues (Insulin Glargine and Insulin Aspart) in Insulin naïve Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-4157; 2014-003708-62 (EudraCT Number); U1111-1158-7280 (Other: WHO)
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2018-09

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIAsp (Experimental)
  Interventions: Drug: biphasic insulin aspart 30
- IGlar + IAsp (Active Comparator)
  Interventions: Drug: insulin glargine; Drug: insulin aspart

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Injected s.c./subcutaneously once daily with the largest meal Subjects should continue their pre-trial metformin and sulfonylurea dosages all throughout the trial while other oral antidiabetic drugs will be discontinued.
  Arms: BIAsp
Drug: insulin glargine — Injected s.c./subcutaneously once daily at the same time every day, with the possibility of treatment intensification with insulin aspart (Basal-bolus arm) Subjects should continue their pre-trial metformin and sulfonylurea dosages all throughout the trial while other oral antidiabetic drugs will be discontinued.
  Arms: IGlar + IAsp
Drug: insulin aspart — Injected s.c./subcutaneously once daily.
  Arms: IGlar + IAsp

SUMMARY:
This trial is conducted globally. The aim of this trial is to compare stepwise insulin intensification of biphasic insulin aspart (BIAsp) 30 and basal-bolus therapy with insulin glargine and insulin aspart in insulin naïve type 2 diabetic patients inadequately controlled on oral anti-diabetic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male or female, age at least 18 years at the time of signing informed consent
* Type 2 diabetes subjects clinically diagnosed at least 6 months prior to screening
* Treatment with stable daily dose (for at least 90 days prior to screening) of: - Metformin (equal or above 1000 mg or maximum tolerated dose documented in the patient medical record) and - Sulfonylurea - and willing to discontinue any other oral antidiabetic drugs containing insulin secretagogues, DPP4i (dipeptidyl peptidase-4 inhibitor), SGLT2 (sodium glucose co-transporter 2), colesevelam, bromocriptin and/or combination products at randomisation
* Insulin-naïve. Short term insulin treatment for acute illnesses for a total of 14 days or less is allowed as is prior insulin treatment for gestational diabetes
* HbA1c (glycosylated haemoglobin) 7.0-9.5 % (both inclusive) analysed by central laboratory
* Willing to consume 3 main meals daily (morning, mid-day and evening) throughout the entire trial. The definition for 'main meal' will be according to the investigator's discretion

Exclusion Criteria:

* Anticipated initiation or change in concomitant medications known to affect weight or glucose metabolism, in excess of 14 days (i.e. sibutramine, orlistat, thyroid hormones, systemic corticosteroids and other weight loss/modifying agents)
* Impaired liver function, defined as ALT (alanine aminotransferase) at least 2.5 times upper limit of normal (central laboratory value measured at screening visit)
* Inadequately treated high blood pressure defined as Class 2 hypertension or higher (i.e. systolic blood pressure equal to or above 160 mm Hg or diastolic equal to or above 100 mm Hg) in accordance with the National High Blood Pressure Education Program, 7th Joint National Committee1 and ESH/ESC 2013 Guidelines2
* Within the past 180 days prior to randomisation, any of the following: Myocardial Infarction, stroke or hospitalization for unstable angina and /or transient ischemic attack

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2016-09-20 (Actual); Study Completion 2016-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (31):
- Australia (5):
  - Novo Nordisk Investigational Site, Broadmeadow, New South Wales
  - Novo Nordisk Investigational Site, Coffs Harbour, New South Wales
  - Novo Nordisk Investigational Site, Ipswich, Queensland
  - Novo Nordisk Investigational Site, Fitzroy, Victoria
  - Novo Nordisk Investigational Site, Melbourne, Victoria
- Bulgaria (3):
  - Novo Nordisk Investigational Site, Petrich
  - Novo Nordisk Investigational Site, Sliven
  - Novo Nordisk Investigational Site, Sofia
- Hungary (2):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Nyíregyhaza
- India (7):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Madurai, Tamil Nadu
  - Novo Nordisk Investigational Site, Vellore, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, New Delhi
- Serbia (2):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Niš
- Novo Nordisk Investigational Site, Seoul, South Korea
- Thailand (3):
  - Novo Nordisk Investigational Site, Bangkok
  - Novo Nordisk Investigational Site, Bangkoknoi, Bangkok
  - Novo Nordisk Investigational Site, Khon Kaen
- Turkey (Türkiye) (4):
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Malatya
  - Novo Nordisk Investigational Site, Rize
- United Arab Emirates (4):
  - Novo Nordisk Investigational Site, Ajman
  - Novo Nordisk Investigational Site, Dubai
  - Novo Nordisk Investigational Site, Ras al-Khaimah
  - Novo Nordisk Investigational Site, Umm Al Quwain City

REFERENCES:
- [Result] Linjawi S, Lee BW, Tabak O, Lovdahl S, Werther S, Abusnana S. A 32-Week Randomized Comparison of Stepwise Insulin Intensification of Biphasic Insulin Aspart (BIAsp 30) Versus Basal-Bolus Therapy in Insulin-Naive Patients with Type 2 Diabetes. Diabetes Ther. 2018 Feb;9(1):1-11. doi: 10.1007/s13300-017-0334-8. Epub 2017 Nov 11. PMID 29129018
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 41 sites in 9 countries, as follows: Australia: 4 sites; Bulgaria: 5 sites; Hungary: 3 sites; India: 7 sites; Korea, Republic of: 4 sites; Serbia: 5 sites; Thailand: 4 sites; Turkey: 5 sites; United Arab Emirates: 4 sites.
Groups:
- BIAsp 30: Subjects received subcutaneous (s.c.) injection of biphasic insulin aspart 30 (BIAsp 30-a mixture of soluble insulin aspart [IAsp] 30% and protaminated IAsp 70%) during a 32-week treatment period (divided into 4 periods of 8 weeks each). Subjects started treatment with 1 daily injection of BIAsp 30 (starting dose 12 unit) with the largest meal. Insulin titration: Subjects underwent weekly insulin dose titration during entire treatment period in order to achieve the pre-meal self-measured plasma glucose (SMPG) target of 4.4-6.1 mmol/L (80-110 mg/dL). Insulin intensification: At the end of each 8-week period, insulin treatment was intensified in stepwise manner by adding an additional injection of BIAsp 30 depending on whether subjects achieved the pre-defined glycaemic target (hemoglobin A1c [HbA1c] <7.0%). Subjects had the possibility of receiving up to 3 daily injections of BIAsp 30. Subjects continued pre-trial treatment with metformin and sulphonylurea (SU) throughout the trial.
- Basal-bolus: Subjects received s.c. injections of insulin glargine (IGlar) during a 32-week treatment period (divided into 4 periods of 8 weeks each). Subjects started with 1 daily injection of IGlar (administrated at same point of time every day) with starting dose of 10 units. Insulin titration: Subjects underwent a weekly insulin dose titration during the entire treatment period in order to achieve the pre-meal SMPG target of 4.4-6.1 mmol/L (80-110 mg/dL). Insulin intensification: At the end of each 8-week period, insulin treatment was intensified in a stepwise manner by adding an additional injection of IAsp depending on whether subjects achieved the pre-defined glycaemic target (HbA1c <7.0%). Subjects had the possibility of receiving 1 daily injection of IGlar plus up to 3 daily injections of IAsp. Subjects continued their pre-trial treatment with metformin and SU throughout the trial.
Period: Overall Study
Arm/Group | BIAsp 30 | Basal-bolus
Started | 168 | 167
Exposed | 166 | 166
Completed | 149 | 155
Not Completed | 19 | 12
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 7 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 8 | 4
Not completed — Unclassified | 4 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomised subjects.
Groups:
- BIAsp 30: Subjects received s.c. injection of BIAsp 30 (a mixture of soluble IAsp 30% and protaminated IAsp 70%) during a 32-week treatment period (divided into 4 periods of 8 weeks each). Subjects started treatment with 1 daily injection of BIAsp 30 (starting dose 12 unit) with the largest meal. Insulin titration: Subjects underwent weekly insulin dose titration during entire treatment period in order to achieve the pre-meal SMPG target of 4.4-6.1 mmol/L (80-110 mg/dL). Insulin intensification: At the end of each 8-week period, insulin treatment was intensified in stepwise manner by adding an additional injection of BIAsp 30 depending on whether subjects achieved the pre-defined glycaemic target (HbA1c <7.0%). Subjects had the possibility of receiving up to 3 daily injections of BIAsp 30. Subjects continued pre-trial treatment with metformin and SU throughout the trial.
- Basal-bolus: Subjects received s.c. injections of IGlar during a 32-week treatment period (divided into 4 periods of 8 weeks each). Subjects started with 1 daily injection of IGlar (administrated at same point of time every day) with starting dose of 10 units. Insulin titration: Subjects underwent a weekly insulin dose titration during the entire treatment period in order to achieve the pre-meal SMPG target of 4.4-6.1 mmol/L (80-110 mg/dL). Insulin intensification: At the end of each 8-week period, insulin treatment was intensified in a stepwise manner by adding an additional injection of IAsp depending on whether subjects achieved the pre-defined glycaemic target (HbA1c <7.0%). Subjects had the possibility of receiving 1 daily injection of IGlar plus up to 3 daily injections of IAsp. Subjects continued their pre-trial treatment with metformin and SU throughout the trial.
- Total: Total of all reporting groups
Arm/Group | BIAsp 30 | Basal-bolus | Total
Number analyzed (Participants) | 168 | 167 | 335
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (10.4) | 56.5 (10.1) | 56.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 90 | 169
  Male | 89 | 77 | 166
HbA1c [Mean (Standard Deviation); unit: Percentage of HbA1c] | 8.31 (0.73) | 8.23 (0.69) | 8.27 (0.71)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Glycosylated Haemoglobin)
Description: Change in HbA1c from baseline (week 0) to week 32.
Time Frame: Week 0, week 32
Population: Full analysis set. Week 32 data are presented after application of Last observation carried forward; 164 subjects contributed in each arm.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | BIAsp 30 | Basal-bolus
Number analyzed (Participants) | 164 | 164
Percentage of HbA1c | -1.16 (0.98) | -1.30 (0.90)
Statistical Analysis 1: Comparison: BIAsp 30 vs Basal-bolus; Analysis was performed using mixed model repeated measurements including treatment, region, and strata as fixed effects, HbA1c at baseline as covariate, interactions between all fixed effects and visit and using an unstructured residual covariance matrix; Test type: Superiority or Other; p = 0.0435, Mixed Models Analysis; Treatment difference at week 32 = 0.18, 95% CI 2-sided [0.01 to 0.36] — 'Treatment difference' refers to "BIAsp 30 minus Basal-bolus

2. Secondary Outcome: HbA1c Below 7.0% Without Severe Hypoglycaemic Episodes
Description: Percentage of subjects with HbA1c below 7.0% after 32 weeks of randomised treatment without treatment emergent severe hypoglycaemic episodes during the last 12 weeks of treatment. Subjects withdrawn before 32 weeks were handled as non-responders. Severe hypoglycaemic episode was defined as an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose (PG) concentrations may not be available during an event, but neurological recovery following the return of PG to normal is considered sufficient evidence that the event was induced by a low PG concentration.
Time Frame: After 32 weeks of treatment (yes/no)
Population: Full analysis set.
Measure: Number; unit: Percentage of subjects
Arm/Group | BIAsp 30 | Basal-bolus
Number analyzed (Participants) | 168 | 167
Percentage of subjects
  Yes | 42.3 | 56.3
  No | 57.7 | 43.7

3. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes Classified According to the American Diabetes Association (ADA) and the Novo Nordisk Definitions
Description: Hypoglycaemic episodes were classified as severe, Asymptomatic, Documented symptomatic, Pseudo, and Probable symptomatic as per ADA classification. As symptoms of hypoglycaemia occur below a PG level of 3.1 mmol/L, (56 mg/dL) Novo Nordisk classification included hypoglycaemia with plasma glucose (PG) levels below 3.1 mmol/L (56 mg/dL) in the definition of blood glucose confirmed hypoglycaemia. Hence, Novo Nordisk classification included following types of hypoglycaemia in addition to ADA classification: Severe hypoglycaemia, Symptomatic blood glucose confirmed hypoglycaemia, Asymptomatic blood glucose confirmed hypoglycaemia, Severe or blood glucose confirmed symptomatic hypoglycaemia, Blood glucose confirmed hypoglycaemia, and Severe or blood glucose confirmed hypoglycaemia. Reported data represents total of all hypoglycaemic episodes.
Time Frame: Weeks 0-32
Population: The safety analysis set included all subjects receiving at least one dose of the investigational product or its comparator.
Measure: Number; unit: Hypoglycaemic episodes
Arm/Group | BIAsp 30 | Basal-bolus
Number analyzed (Participants) | 166 | 166
Hypoglycaemic episodes
  ADA classification | 1650 | 1841
  Novo Nordisk classification | 1650 | 1841

4. Secondary Outcome: Total Daily Insulin Dose
Description: Total daily insulin dose in the basal bolus treatment group and in BIAsp 30 treatment group at each week of each treatment.
Time Frame: Weeks 0-32
Population: Safety analysis set. Number analysed=number of subjects with available data for individual timepoints.
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | BIAsp 30 | Basal-bolus
Number analyzed (Participants) | 166 | 166
U/kg
  Week 1: number analyzed (Participants) | 164 | 165
  Week 1 | 0.157 (0.038) | 0.127 (0.026)
  Week 2: number analyzed (Participants) | 162 | 165
  Week 2 | 0.187 (0.053) | 0.167 (0.042)
  Week 3: number analyzed (Participants) | 163 | 164
  Week 3 | 0.214 (0.070) | 0.197 (0.061)
  Week 4: number analyzed (Participants) | 160 | 161
  Week 4 | 0.238 (0.088) | 0.224 (0.076)
  Week 5: number analyzed (Participants) | 158 | 158
  Week 5 | 0.259 (0.102) | 0.244 (0.088)
  Week 6: number analyzed (Participants) | 157 | 161
  Week 6 | 0.280 (0.114) | 0.264 (0.100)
  Week 7: number analyzed (Participants) | 155 | 161
  Week 7 | 0.296 (0.131) | 0.281 (0.110)
  Week 8: number analyzed (Participants) | 155 | 161
  Week 8 | 0.308 (0.145) | 0.296 (0.119)
  Week 9: number analyzed (Participants) | 154 | 159
  Week 9 | 0.369 (0.172) | 0.339 (0.137)
  Week 10: number analyzed (Participants) | 154 | 159
  Week 10 | 0.397 (0.199) | 0.365 (0.160)
  Week 11: number analyzed (Participants) | 154 | 159
  Week 11 | 0.421 (0.224) | 0.391 (0.182)
  Week 12: number analyzed (Participants) | 153 | 160
  Week 12 | 0.443 (0.245) | 0.413 (0.202)
  Week 13: number analyzed (Participants) | 150 | 158
  Week 13 | 0.456 (0.267) | 0.425 (0.214)
  Week 14: number analyzed (Participants) | 151 | 158
  Week 14 | 0.472 (0.277) | 0.439 (0.228)
  Week 15: number analyzed (Participants) | 151 | 159
  Week 15 | 0.487 (0.295) | 0.455 (0.237)
  Week 16: number analyzed (Participants) | 151 | 159
  Week 16 | 0.501 (0.308) | 0.468 (0.248)
  Week 17: number analyzed (Participants) | 149 | 156
  Week 17 | 0.528 (0.324) | 0.496 (0.270)
  Week 18: number analyzed (Participants) | 150 | 157
  Week 18 | 0.546 (0.334) | 0.516 (0.294)
  Week 19: number analyzed (Participants) | 149 | 157
  Week 19 | 0.557 (0.353) | 0.532 (0.316)
  Week 20: number analyzed (Participants) | 148 | 155
  Week 20 | 0.569 (0.367) | 0.544 (0.320)
  Week 21: number analyzed (Participants) | 149 | 155
  Week 21 | 0.588 (0.387) | 0.563 (0.347)
  Week 22: number analyzed (Participants) | 149 | 156
  Week 22 | 0.602 (0.401) | 0.580 (0.359)
  Week 23: number analyzed (Participants) | 148 | 156
  Week 23 | 0.607 (0.411) | 0.590 (0.373)
  Week 24: number analyzed (Participants) | 148 | 156
  Week 24 | 0.615 (0.426) | 0.605 (0.386)
  Week 25: number analyzed (Participants) | 147 | 154
  Week 25 | 0.628 (0.435) | 0.618 (0.398)
  Week 26: number analyzed (Participants) | 147 | 156
  Week 26 | 0.643 (0.454) | 0.643 (0.434)
  Week 27: number analyzed (Participants) | 149 | 155
  Week 27 | 0.661 (0.472) | 0.653 (0.452)
  Week 28: number analyzed (Participants) | 149 | 155
  Week 28 | 0.671 (0.487) | 0.664 (0.466)
  Week 29: number analyzed (Participants) | 149 | 155
  Week 29 | 0.688 (0.509) | 0.674 (0.484)
  Week 30: number analyzed (Participants) | 149 | 155
  Week 30 | 0.692 (0.511) | 0.682 (0.497)
  Week 31: number analyzed (Participants) | 149 | 155
  Week 31 | 0.703 (0.525) | 0.693 (0.515)
  Week 32: number analyzed (Participants) | 153 | 155
  Week 32 | 0.700 (0.542) | 0.708 (0.537)

ADVERSE EVENTS:
Time Frame: From first randomised treatment (week 0) to last randomised treatment (week 32) + 7 days.
Description: The safety analysis set included all subjects receiving at least one dose of the investigational product or its comparator. All adverse events mentioned here were treatment emergent (an event that has an onset date on or after the first day of exposure to randomised treatment, and no later than 7 days after the last day of randomised treatment).
Arm/Group | BIAsp 30 | Basal-bolus
Serious Adverse Events (participants affected / at risk) | 14/166 | 12/166
Other Adverse Events (participants affected / at risk) | 37/166 | 40/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIAsp 30 (N=166) | Basal-bolus (N=166)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 3 (8)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 2 (3)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIAsp 30 (N=166) | Basal-bolus (N=166)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (16) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (13) | 8 (9)
Diarrhoea (Gastrointestinal disorders) | 10 (19) | 11 (12)
Headache (Nervous system disorders) | 12 (24) | 15 (27)
Nasopharyngitis (Infections and infestations) | 21 (31) | 18 (27)
Upper respiratory tract infection (Infections and infestations) | 11 (15) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.